CLINICAL TRIAL: NCT06277752
Title: A Randomized, Open-label,Single Dosing Clinical Trail to Investigate the Pharmacokinetic/Pharmacodynamic Characteristics of IBI128 in Chinese Healthy Subjects
Brief Title: A Study to Investigate the Pharmacokinetic/Pharmacodynamic Characteristics of IBI128(A New Xanthine Oxidase Inhibitor)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI128A101
Record Dates: First submitted 2024-02-04; First posted 2024-02-26 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Gout Arthritis
MeSH Terms: conditions — Arthritis, Gouty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI128 (Experimental): IBI128 po. QD(Quaque Die)
  Interventions: Drug: dose-5 group; Drug: dose-1 group; Drug: dose-2 group; Drug: dose-4 group; Drug: dose-3 group

INTERVENTIONS:
Drug: dose-5 group — IBI128 300mg po. QD(Quaque Die)
Drug: dose-1 group — IBI128 25mg po. QD(Quaque Die)
Drug: dose-2 group — IBI128 50mg po. QD(Quaque Die)
Drug: dose-4 group — IBI128 200mg po. QD(Quaque Die)
Drug: dose-3 group — IBI128 100mg po. QD(Quaque Die)

SUMMARY:
A Phase I study to evaluate the pharmacokinetic/pharmacodynamic characteristics,safety and tolerability of IBI128 after multidosing in Chinese health subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 50 years at screening;
2. Subjects with a Body Mass Index (BMI) between 18.0 (inclusive) and 28.0 kg/m2 (inclusive); and a total body weight ≥55kg (male） and 45kg (female)
3. Participants who are overtly healthy as determined by medical evaluation including medical history, laboratory tests, vital signs and standard 12 lead ECGs.
4. Subject is willing to participate and to Sign written informed consent form.

Exclusion Criteria:

1. Subjects with a history of hypersensitivities to investigational products, including drug allergies (caused by aspirin, antibiotics, etc.), or a history of clinically significant hypersensitivities
2. Subjects with evidence or a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or surgery (except simple appendectomy or repair of hernia) that may influence drug absorption
3. Subjects with evidence or a history of clinically significant hepatic (including carrier of viral hepatitis), renal, neurologic, immunologic, pulmonary, endocrine, hematological, neoplastic, cardiovascular or psychiatric (mood disorder, obsessive-compulsive disorder, etc.) diseases.
4. Subjects with a history or current have mental disease.
5. Subjects who have taken any medicine that may affect outcomes within 30 days before the first administration of the investigational product.
6. Subject who have taken IBI128 in other studies.
7. Subjects who have a history of acute arthiritis.
8. Pregnant women or breast-feeding women or men and women who has possibility of pregnancy.
9. Subjects judged not eligible for the study after reviewing the clinical laboratory results or other reasons by the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
PK parameter: Cmax | Up to Day 8
  Maximum plasma concentration(Cmax) of IBI128
PK parameter: AUC | Up to Day 8
  Area under the concentration-time curve （AUC）of IBI128
PK parameter: Tmax | Up to Day 8
  Time to ahieve Cmax
PK parameter: T1/2 | Up to Day 8
  The time that takes for the dlimination processes to reduce the plasma concentration of the drug in the body by 50%.

SECONDARY OUTCOMES:
Safety parameter: AE | Up to Day 8
  Number of subjects with Adverse Event
PD parameter: serum UA (uric acid） | Up to Day 8
  The Percentage change of serum UA assesed by Area Under Curve 24，Cmean,24，Cmean,24 of IBI128 from baseline.
Tolerability parameter: SAE | Up to Day 8
  Number of subjects with Serious Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated, Zhengzhou, Henan, China